CLINICAL TRIAL: NCT03131947
Title: HOST Study - HIV in Orthopaedic Skeletal Trauma Study; Fracture Healing in HIV-positive Patients
Brief Title: HIV in Orthopaedic Skeletal Trauma Study
Acronym: HOST
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Wellcome Trust Liverpool Glasgow Centre for Global Health Research (Other)
Collaborators: Professor David Lalloo (Unknown); Professor Hamish Simpson (Unknown); Professor William J Harrison (Unknown); Professor Sithombo Maqungo (Unknown)
Responsible Party: Principal Investigator, John Spafford, Wellcome Trust Clinical Research and Training Fellow, Wellcome Trust Liverpool Glasgow Centre for Global Health Research
Other Study IDs: HOST STUDY
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2018-05-22 (Actual); Status verified 2018-05

CONDITIONS: Fracture Healing in HIV-positive Patients

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Union: Radiological union on RUST score (figure 2) (score of 3 on at least 3 cortices in AP, lateral, medial or posterior cortex - total of 9 or more) within 6 months of surgery
  Interventions: Other: HIV positive patients
- Delayed union: Impaired bone healing at six months (RUST score < 9)
  Interventions: Other: HIV positive patients

INTERVENTIONS:
Other: HIV positive patients — As above
  Other Names: No intervention, patients undergo standard surgery for their fracture management.

SUMMARY:
Adult patients > 18 years with fresh (within 2 weeks of injury), closed and open, tibia and femur fractures who undergo IM nailing for fracture fixation will be eligible for the study. Participants will be recruited over 24 months. Participants will undergo a baseline questionnaire, HIV testing and assessment of their BMD. They will be followed up at 6 weeks, and 3, 6 and 12 months. All adult patients who develop delayed bone union at 6 month follow up will be considered cases. Adult patients who show evidence of radiological union at 6 months or less will be considered controls.

DETAILED DESCRIPTION:
1. Primary research question Does Human Immunodeficiency Virus (HIV) alter the fracture repair process?
2. Aim To establish whether HIV is a risk factor for the development of delayed bone union or nonunion following a fracture.
3. Study

   1. Setting Orthopaedic and Trauma Department, Groote Schuur Hospital (GSH), Cape Town, South Africa.
   2. Study design Case-cohort study of patients undergoing fracture surgery at GSH, Cape Town, South Africa.
   3. Study population Adult patients > 18 years with fresh (within 2 weeks of injury), closed and open, tibia and femur fractures who undergo intramedullary (IM) nailing for fracture fixation.
   4. Study summary Adult patients > 18 years with fresh (within 2 weeks of injury), closed and open, tibia and femur fractures who undergo intramedullary (IM) nailing for fracture fixation will be potentially eligible for inclusion in the study. Participants will undergo a baseline questionnaire, assessment of their HIV status and measurement of their bone mineral density (BMD) using a Dual Energy X-ray Absorbometry (DEXA) Heel Scanner.

Participants will be followed up at 2 weeks, and 3, 6 and 12 months. X-rays will be performed at 3, 6 and 12 months. Bone healing will be assessed using a validated X-ray scoring system - the Radiological Union Scoring system for the Tibia (RUST scoring system).(19), (20) An independent observer blinded to HIV status will assess radiological fracture union. Participants will be recruited over 24 months.

All adult patients treated at GSH with IM nailing of the tibia or femur and develop delayed bone union at 6 month follow up will be considered cases. Adult patients who show evidence of radiological union at 6 months or less will be considered controls.

ELIGIBILITY:
Inclusion criteria;

* They are older than 18 years old
* Present to the GSH within 2 weeks of injury
* Sustained a closed or open fracture of tibia and femur fractures
* Undergo IM nailing for fracture fixation

Exclusion Criteria:

* Major head injury
* Pre-surgical infection at the fracture site
* Open injury for >48 hours before the first debridement.
* Severe burns
* Pathological fracture
* There is evidence that the patient would be unable to adhere to study procedures, complete questionnaires or attend follow up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients > 18 years with fresh (within 2 weeks of injury), closed and open, tibia and femur fractures who undergo intramedullary (IM) nailing for fracture fixation will be potentially eligible for inclusion in the study.
Sampling Method: Non-Probability Sample
Enrollment: 420 (Estimated)
Dates: Start 2017-09-28 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Delayed fracture healing | 6 months
  Incidence of delayed bone union in patients treated at GSH in HIV positive and negative patients

SECONDARY OUTCOMES:
Nonunion | 12 months
  Incidence of nonunion in patients treated at GSH in HIV positive and negative patients
Infection | 12 months
  Incidence of superficial, deep and late wound infections in patients treated at GSH in HIV positive and negative patients

CONTACTS AND LOCATIONS:
Locations (1):
- Groote Schuur Hospital, Cape Town, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Graham SM, Maqungo S, Laubscher M, Ferreira N, Held M, Harrison WJ, Simpson AH, MacPherson P, Lalloo DG. Fracture Healing in Patients With HIV in South Africa: A Prospective Cohort Study. J Acquir Immune Defic Syndr. 2021 Aug 15;87(5):1214-1220. doi: 10.1097/QAI.0000000000002720. PMID 33990496